CLINICAL TRIAL: NCT06967675
Title: Changes in Perfusion Index Under Low-Flow Anesthesia and Its Effects on Postoperative Emergence in Pediatric Patients
Brief Title: Perfusion Index in Pediatric Low-Flow Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: haseki low flow
Record Dates: First submitted 2025-05-03; First posted 2025-05-13 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Perfusion Index; Low-Flow Anesthesia; Postoperative Recovery

STUDY DESIGN:
Intervention Model Description: ediatric patients undergoing elective surgery will be followed in two naturally assigned groups based on anesthesia flow rate: low-flow (LFA) and normal-flow (HFA). No intervention will be applied outside routine clinical care, and all data will be collected through perioperative monitoring.
Who Masked: Participant, Investigator
Masking Description: Group allocation is determined by the anesthesia provider during routine care. Both the participant and the outcome assessor are blinded to group assignment. Data analysis is performed without group identifiers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Flow Anesthesia Group (LFA) (Experimental): Patients will receive general anesthesia using a fresh gas flow rate of 1 L/min (50% O₂ + 50% air). Perfusion index and hemodynamic parameters will be monitored at predetermined time points.
  Interventions: Procedure: Low-Flow Anesthesia (LFA)
- Normal-Flow Anesthesia Group (HFA) (Active Comparator): Patients will receive general anesthesia using a fresh gas flow rate of 2 L/min (50% O₂ + 50% air). Perfusion index and hemodynamic parameters will be monitored at the same time points.
  Interventions: Procedure: Low-Flow Anesthesia (LFA)

INTERVENTIONS:
Procedure: Low-Flow Anesthesia (LFA) — General anesthesia with a fresh gas flow rate of 1 L/min (50% oxygen + 50% air).

SUMMARY:
This study aims to evaluate changes in perfusion index (PI) in pediatric patients undergoing elective surgery under low-flow anesthesia. PI will be monitored at multiple intraoperative and postoperative time points to assess its relationship with hemodynamic stability and depth of anesthesia. The study will also investigate whether low-flow anesthesia affects the incidence of emergence agitation (EA). Patients will be assigned to either low-flow or normal-flow anesthesia groups based on routine clinical practice. No intervention will be applied beyond standard care. The findings are expected to provide insight into the predictive value of PI in postoperative recovery and support safer anesthesia practices in pediatric populations.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II pediatric patients
* Age 2 to 12 years
* Undergoing elective surgery lasting between 1-6 hours
* Informed consent obtained from parents/guardians

Exclusion Criteria:

* Cardiovascular, respiratory, neurological, metabolic, or endocrine disorders
* Premature birth with corrected age < 2 years
* Obesity or severe malnutrition (BMI <5th or >95th percentile)
* Psychiatric or neurodevelopmental disorders (e.g., autism)
* Malignant hyperthermia or hypersensitivity to anesthetics
* Emergency surgeries
* Lack of IV access requiring inhalational induction
* Contraindications to low-flow anesthesia including:
* Severe pulmonary disease
* Congenital heart disease with shunt physiology
* Anticipated high oxygen demand
* Airway obstruction risk
* Surgeries requiring high gas flow or >6 hours duration

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Change in Perfusion Index (PI) | From induction to 30 minutes after extubation
  Perfusion Index (PI) will be measured at 11 predefined perioperative time points to assess its intraoperative variation and its potential correlation with anesthesia depth and emergence profile in pediatric patients undergoing low-flow vs normal-flow anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krishnamohan A, Siriwardana V, Skowno JJ. Using a pulse oximeter to determine clinical depth of anesthesia-investigation of the utility of the perfusion index. Paediatr Anaesth. 2016 Nov;26(11):1106-1111. doi: 10.1111/pan.13000. Epub 2016 Aug 28. PMID 27569026
- [Result] RYALINO, CHRISTOPHER, et al. Low-flow anesthesia technique reduces emergence agitation in pediatric patients underwent general anesthesia. Asian Journal of Pharmaceutical and Clinical Research, 2019, 12.5: 139-41.
- [Result] Kowalczyk M, Fijalkowska A, Nestorowicz A. New generation pulse oximetry in the assessment of peripheral perfusion during general anaesthesia - a comparison between propofol and desflurane. Anaesthesiol Intensive Ther. 2013 Jul-Sep;45(3):138-44. doi: 10.5603/AIT.2013.0029. PMID 24092509